CLINICAL TRIAL: NCT05779995
Title: Randomized, Double-blind, Placebo-controlled Phase Ib/Ⅱa Study to Evaluate the Safety, Tolerability, Efficacy, Pharmacokinetics, and Immunogenicity of XW001 Inhalation in Children With Respiratory Syncytial Virus (RSV) Infection in China
Brief Title: A Study To Evaluate the Safety of XW001 Inhalation in Children With RSV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hangzhou Sciwind Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCW1201-3021
Record Dates: First submitted 2023-02-06; First posted 2023-03-22 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2023-07

CONDITIONS: RSV Infection
Keywords: XW001; Respiratory Syncytial Virus
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — XW001

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- C1-XW001 (Experimental): Low dose of XW001 once daily
  Interventions: Drug: XW001
- C1-Placebo (Placebo Comparator): Matched Placebo once daily
  Interventions: Drug: Placebo
- C2-XW001 (Experimental): Medium dose of XW001 once daily
  Interventions: Drug: XW001
- C2-Placebo (Placebo Comparator): Matched Placebo once daily
  Interventions: Drug: Placebo
- C3-XW001 (Experimental): High dose of XW001 once daily
  Interventions: Drug: XW001
- C3-Placebo (Placebo Comparator): Matched Placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XW001 — Inhalation solution
  Arms: C1-XW001; C2-XW001; C3-XW001
Drug: Placebo — Inhalation solution with matched volume
  Arms: C1-Placebo; C2-Placebo; C3-Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled Phase Ib/IIa study to evaluate the safety, tolerability, efficacy, pharmacokinetics, and immunogenicity of XW001 inhalation in children with RSV infection in China

DETAILED DESCRIPTION:
In this study, eligible participants will be randomized in a 4:1 ratio to receive XW001 inhalation (one of three dosage groups) or placebo once a day for 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 1 to 24 months (inclusive) at screening;
2. Weight: 3-20 kg, inclusive;
3. Positive RSV test within 36 hours before randomization;
4. Symptomatic at screening and randomization, and the onset of RSV symptoms is within 5 days prior to the first dose of XW001;
5. Parents/legal guardians are able to understand the purpose and procedures of the study, and are able to provide informed consent.

Exclusion Criteria:

1. Immunocompromised as determined by the investigator;
2. Known to have undergone or planned for bone marrow, stem cells, or other organ transplants, or are currently on immunosuppressive treatment;
3. Positive for HBV, HCV or HIV, or patient <6 months old whose mother is positive for HIV;
4. History of seizures or epilepsy, including febrile seizure;
5. Known to have received any prohibited medications defined by the protocol within 3 days prior to randomization;
6. History of any surgery within 30 days prior to randomization;
7. Severe dental or facial deformity that will impact on usage of nebulizer;
8. History of receiving measles, mumps, rubella or other vaccines within 7 days prior to screening;
9. Known to have received any investigational medicinal products or devices in the past 30 days;
10. Any other underlying conditions that make the patient unlikely to complete the study in the opinion of the investigator.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events after receiving XW001 | Day 1 to Day 28

SECONDARY OUTCOMES:
Change from baseline in RSV load via nasopharyngeal swab | Baseline, Day 2 to Day 8
Change from baseline in Wang Respiratory Score | Baseline, Day 2 to Day 8
Pharmacokinetics-Plasma level of XW001 | Baseline, Day 8
Immunogenicity-Anti-drug Antibody of XW001 | Baseline, Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Hanmin Liu, Dr, Principal Investigator — West China Second University Hospital; Qin Yu, Principal Investigator — West China Second University Hospital
Locations (1):
- West China Second University Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No